CLINICAL TRIAL: NCT06281171
Title: SkillTalk: Using Streaming Video for Young Adults With Autism Spectrum Disorder to Build Microskills to Develop and Sustain Relationships for Healthy and Independent Living Spectrum Disorder
Brief Title: Evaluation of SkillTalk for Autistic Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dfusion Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 90BISB0022
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; Autism; Microskills; Video Training; Communication Skills; Young Adult
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Library Group (Experimental): This arm will receive the intervention. This intervention is access to the SkillTalk for AYA Microskills video library, about 60 minutes in duration. The library includes a curriculum covering skills such as setting boundaries, resolving conflict, and emotional regulation.
  Interventions: Other: SkillTalk for Autistic Young Adults
- Flyer Library Group (Active Comparator): During the intervention period, arm 2 will receive flyers with information on relationship skills. This arm will receive the intervention upon completion of follow-up study activities.
  Interventions: Other: Flyer Library

INTERVENTIONS:
Other: SkillTalk for Autistic Young Adults — A Microskills video training library on communication skills for autistic young adults.
  Arms: Video Library Group
Other: Flyer Library — A collection of existing online resources on relationship skills
  Arms: Flyer Library Group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of using a Microskills video training library for young adults, aged 18-28, with autism spectrum disorder (ASD) to enhance their skills in developing and maintaining healthy relationships.

The main questions it aims to answer are:

* Does using SkillTalk increase autistic young adults skills in the communications skills that are demonstrated in the video curriculum (skills: resolve conflict, compromise, give feedback)?
* Does using SkillTalk increase reported confidence and satisfaction in communication and relationship skills?
* Does using SkillTalk increase interpersonal competence?
* Does using SkillTalk increase ability to cope with rejection?
* Does using SkillTalk improve mental health and wellbeing?

Participants will be asked to:

* Take a survey at the beginning of the study, after one month the end of the study, and at 3-month follow up
* Participate in recorded video calls with projects staff, comprised of 2-3 brief roleplay scenarios of relationship skills at the beginning of the study, after one month the end of the study, and at 3-month follow up
* Watch a minimum of 85% of the 60 minutes of video assigned

DETAILED DESCRIPTION:
The proposed project will establish the efficacy of using SkillTalk for Autistic Young Adults online video library to improve the relationship and communication skills of young adults on the autism spectrum. A randomized controlled trial is being conducted to assess the impact of the resource on participant skill demonstration and confidence, interpersonal competence, mental health and wellbeing. Participants will be young adults, aged 18-28, have ASD, with reciprocal communication skills and receptive language skills. Participants with diagnosed intellectual disabilities will be excluded from the study.

Participants are primarily being recruited with assistance from agencies/organizations that serve those with ASD, community and professional advisory board members, and other community networks. It is also likely that participants will refer other autistic young adults participation.

The study design will be a randomized controlled trial with pre- and post-assessment, and a 3-month follow-up assessment (4 months after start of study), each including a survey and a facilitated roleplay via video call. After completing the baseline activities, half (55) of the participants will be randomly assigned to the SkillTalk AYA intervention group which will receive access to the SkillTalk AYA web site. The control group will receive written materials with similar content. For baseline, participants will take a survey and take part in a brief facilitated role play of 3 simple relationship scenarios, one on one with a project staff member. Intervention participants will have access to SkillTalk AYA for 1 month. At the conclusion of the month period, they will participate in an immediate post-test which will again include a survey and a facilitated role play session. Three months after the conclusion of the access period participants will take a survey and take part in a final role play session. At the conclusion of the 4-month period the control group participants will be provided with access to the SkillTalk AYA materials.

ELIGIBILITY:
Inclusion Criteria:

* young adults, aged 18-28
* have ASD, with
* reciprocal communication skills and receptive language skills.

Eligibility will be determined by study staff with screener questions posed to the participants about their age, ASD status (self-report based on self-determination), and comfort with the study activities.

Exclusion Criteria:

- Interested individuals participate in a consent screening call where they are asked to answer four simple questions about the information provided in the consent form. Participants who are unable to answer these questions correctly after prompting from study staff are excluded from the study.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Regina Firpo-Triplett, MPH, Principal Investigator — dfusion Inc
Locations (1):
- Virtual Study, Santa Cruz, California, United States

IPD SHARING:
Plan to Share IPD: No
The research is being conducted under a Small Business Innovation Grant (SBIR) in support of product development and is considered proprietary to the business.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited via social media advertisement from Jan-Mar, 2024. A post about the study was boosted 3 times on both Instagram and Facebook. Posts included a link and a QR code that directed interested individuals to a webpage with further information about the study: https://dfusion.my.canva.site/. They were then provided with a link to an eligibility screener. Eligible individuals were contacted via text or email and provided with access to webpage to book a time for a consent video call.
Pre-assignment Details: Individuals who consented to participate in the study but did not attend the initial study observation and did not respond to attempts to contact were not assigned to study groups.
  All individuals who completed the timepoint on data collection activities were assigned to study groups.
Groups:
- Video Library Group: This arm received the intervention. Participants were assigned their study group following the collection of the timepoint one observational and survey data. Batches were assigned on a weekly basis using stratified randomization to assign participants to the intervention and control groups. The covariates used for stratification were diagnostic status (self-diagnosed and professionally diagnosed and employment/education status (currently employed or attending school or not).
  Following timepoint 1 data collection, participants assigned to the treatment group were provided access to the SkillTalk for AYA Microskills video library and asked to view 75 minutes of assigned videos. The library includes a curriculum covering skills such as setting boundaries, resolving conflict, and emotional regulation. After a month of access, participants took part in a second round of data collection, which was followed by another three months of passive usage of the assigned resource. The study concluded with a final round of data collection.
- Flyer Library Group: This arm received the intervention upon completion of follow-up study activities. Participants were assigned to their study group following the collection of the timepoint one observational and survey data. Batches were assigned on a weekly basis using stratified randomization to assign participants to the intervention and control groups. The covariates used for stratification were diagnostic status (self-diagnosed and professionally diagnosed and employment/education status (currently employed or attending school or not).
  Following timepoint 1 data collection, participants assigned to the attention control group were provided with one month of access to a flyer site with written content on topics not included in the evaluation. This included seven written flyers on the topics of asking for and receiving consent, autism and law enforcement, autistic burnout, navigating health care, unmasking autism, job interview protocol, and workplace accommodations. After a month of access, participants took part in a second round of data collection, which was followed by another three months of passive usage of the assigned resource. The study concluded with a final round of data collection. After the study was finished, control group participants received three months of access to the intervention, to use if they wished.
Period: Timepoint 1
Arm/Group | Video Library Group | Flyer Library Group
Started | 58 | 57
Completed | 58 | 57
Not Completed | 0 | 0
Period: Timepoint 2
Arm/Group | Video Library Group | Flyer Library Group
Started | 58 | 57
Completed | 52 | 53
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 6 | 4
Period: Timepoint 3
Arm/Group | Video Library Group | Flyer Library Group
Started | 52 | 53
Completed | 52 | 48
Not Completed | 0 | 5
Not completed — Lost to Follow-up | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Video Library Group | Flyer Library Group | Total
Number analyzed (Participants) | 58 | 57 | 115
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.11 (2.71) | 23.21 (2.54) | 22.66 (2.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 28 | 64
  Male | 22 | 29 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 35 | 35 | 70
  More than one race | 7 | 8 | 15
  Unknown or Not Reported | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 51 | 50 | 101
  Unknown or Not Reported | 0 | 0 | 0
Diagnostic Status [Count of Participants; unit: Participants]
  Diagnosed by Healthcare Professional | 42 | 34 | 76
  Self Diagnosed | 16 | 23 | 39
Sexuality [Count of Participants; unit: Participants]
  Straight, heterosexual | 6 | 7 | 13
  Bisexual, pansexual | 19 | 18 | 37
  Gay, lesbian, homosexual | 11 | 5 | 16
  Asexual | 7 | 11 | 18
  Queer | 14 | 16 | 30
  Prefer not to answer | 1 | 0 | 1
Education [Count of Participants; unit: Participants]
  Grades 1 through 11 | 1 | 1 | 2
  Regular high school diploma | 3 | 6 | 9
  GED or alternative credential | 2 | 0 | 2
  Less than 1 year of college | 2 | 7 | 9
  1 or more years of college credit, no degree | 21 | 18 | 39
  Associates degree (AA, AS) | 5 | 4 | 9
  Bachelor's degree (BA, BS) | 19 | 15 | 34
  Master's degree (MA, MS, MSW, MEd, MBA, MEng) | 4 | 5 | 9
  Professional degree beyond bachelor's degree | 0 | 0 | 0
  Doctorate degree (PhD, ScD, EdD) | 1 | 1 | 2
Employment Status [Count of Participants; unit: Participants]
  No - but currently looking for a position | 14 | 15 | 29
  No - and not currently looking ofr a position | 6 | 4 | 10
  Yes - full-time | 12 | 16 | 28
  Yes - part-time | 26 | 21 | 47
  Prefer not to answer | 0 | 1 | 1
Housing Situation [Count of Participants; unit: Participants]
  Parent or Guardian | 21 | 25 | 46
  Family | 1 | 1 | 2
  Independently (House or Apartment) | 35 | 30 | 65
  Public Housing | 0 | 1 | 1
  Prefer Not to Answer | 1 | 0 | 1
Relationship Status [Count of Participants; unit: Participants]
  Not currently seeing anyone - but interested | 13 | 12 | 25
  Not currently seeing anyone - and not interested | 7 | 7 | 14
  Casually dating, or hooking up | 12 | 7 | 19
  In a committed long-term partnership or married | 25 | 29 | 54
  Prefer not to answer | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Demonstrated Skill Score in Communication Skills.
Description: Based on a rubric created for this study of the demonstrable skills for the given recorded roleplay conversation. The points earned on the rubric are summed to create a total score. The scale ranges from 0 to 160 with a higher score indicating higher skill usage.
Time Frame: Baseline (T1), 1 month (T2), and 4 months (T3)
Population: All possible participants included at each time point. The reduced numbers reflects those lost to follow up. Further, 3 video files were corrupted or cut off and could not be coded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video Library Group | Flyer Library Group
Number analyzed (Participants) | 58 | 57
score on a scale
  T1 Skill Score: Total All Skills | 72.02 (22.14) | 79.33 (17.76)
  T2 Skill Score: Total All Skills: number analyzed (Participants) | 52 | 54
  T2 Skill Score: Total All Skills | 78.71 (17.60) | 74.65 (18.97)
  T3 Skill Score: Total All Skills: number analyzed (Participants) | 50 | 48
  T3 Skill Score: Total All Skills | 81.04 (14.31) | 81.17 (20.06)
Statistical Analysis 1: Comparison: Video Library Group vs Flyer Library Group; Test type: Superiority; p < .001, Regression, Linear

2. Secondary Outcome: Participant Confidence & Satisfaction in Their Communication Skills
Description: Based on a scale created for the study, the score is comprised of a series of questions about ability to navigate social situations with friends, partners, and acquaintances. The scores from the question are summed to create a total score. The score range is 24 to 120, with higher scores indicating more confidence in ability.
Time Frame: Baseline (T1), 1 month (T2), and 4 months (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video Library Group | Flyer Library Group
Number analyzed (Participants) | 58 | 57
score on a scale
  T3 | 63.01 (10.86) | 63.10 (12.97)
  T2 | 59.15 (11.89) | 59.57 (12.11)
  T1 | 51.07 (11.54) | 53.22 (12.39)
Statistical Analysis 1: Comparison: Video Library Group vs Flyer Library Group; Test type: Superiority; p = .996, t-test, 2 sided

3. Secondary Outcome: Interpersonal Competence Score
Description: Based on the ICQ; Buhrmester et al, 1988. 40-item scale includes subscales: Initiating relationships, self-disclosure, asserting displeasure with others' actions, providing emotional support, and managing interpersonal conflicts. Respondents use a 5-point rating scale to indicate their level of competence and comfort in handling each type of situation (from 1 = "I'm poor at this; I'd feel so uncomfortable and unable to handle this situation, I'd avoid it if possible" to 5 = I'm EXTREMELY good at this; I'd feel very comfortable and could handle this situation very well"). The scores from the question are summed to create a total score. The score range is between 40 and 200. Higher values indicate more communication competence.
Time Frame: Baseline (T1), 1 month (T2), and 4 months (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video Library Group | Flyer Library Group
Number analyzed (Participants) | 58 | 57
score on a scale
  T3 | 137.35 (24.18) | 138.34 (24.95)
  T2 | 126.74 (25.48) | 129.19 (21.81)
  T1 | 113.45 (23.25) | 118.65 (21.46)
Statistical Analysis 1: Comparison: Video Library Group vs Flyer Library Group; Test type: Superiority; p = .782, t-test, 2 sided

4. Secondary Outcome: Coping With Rejection, Jealousy and Relationship Anxiety
Description: Based on a scale by Rothman, Holmes et al 2022. The 16-item scale assessing how participants manage rejection and jealousy. Respondents use a 5-point rating scale to indicate the degree to which they agree with each statement. Add points for each item to create a total scale score. If a respondent skipped two more items, do not score. The score ranges between 16-80. Higher scores indicate better coping with jealousy.
Time Frame: Baseline (T1), 1 month (T2), and 4 months (T3)
Population: All possible participants included at each time point. The reduced numbers reflects those lost to follow-up and individuals who declined to answer specific questions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video Library Group | Flyer Library Group
Number analyzed (Participants) | 58 | 57
score on a scale
  Coping With Rejection Jealousy Scale T1 | 47.60 (10.67) | 47.89 (10.98)
  Coping With Rejection Jealousy Scale T2: number analyzed (Participants) | 52 | 48
  Coping With Rejection Jealousy Scale T2 | 52.58 (10.96) | 51.90 (10.46)
  Coping With Rejection Jealousy Scale T3: number analyzed (Participants) | 51 | 49
  Coping With Rejection Jealousy Scale T3 | 54.88 (10.94) | 55.86 (10.74)
Statistical Analysis 1: Comparison: Video Library Group vs Flyer Library Group; Test type: Superiority; p = 0.54, Regression, Linear

5. Secondary Outcome: PROMIS Depression Scale T-Scores
Description: Patient Reported Outcomes Measurement Information System (PROMIS) Depression Short Form. This adult measure is the 8-item PROMIS Depression Short Form that assesses the pure domain of depression in individuals age 18 and older. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of depression. These raw scores are summed and converted to a T-Score. For the T-Score a higher score indicates greater severity of depression. Generally, a T-score below 55 is considered normal, 55-60 is mild, 60-70 is moderate, and 70 or higher is severe. PROMIS T-scores are standardized to a mean of 50 and a standard deviation of 10.
Time Frame: Baseline (T1), 1 month (T2), and 4 months (T3)
Population: All possible participants included at each time point. The reduced numbers reflects those lost to follow-up and individuals that declined to answer specific survey questions
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Video Library Group | Flyer Library Group
Number analyzed (Participants) | 58 | 57
T-Score
  PROMIS Depression Time 1 | 57.79 (8.79) | 58.64 (7.47)
  PROMIS Depression Time 2: number analyzed (Participants) | 52 | 48
  PROMIS Depression Time 2 | 58.20 (8.28) | 58.30 (8.17)
  PROMIS Depression Time 3: number analyzed (Participants) | 50 | 49
  PROMIS Depression Time 3 | 58.31 (7.46) | 55.36 (9.01)
Statistical Analysis 1: Comparison: Video Library Group vs Flyer Library Group; Test type: Superiority; p = 0.03, Regression, Linear

6. Secondary Outcome: Promise Anxiety Scale
Description: Adult measure is the 7-item PROMIS Anxiety Short Form that assesses the pure domain of anxiety in individuals age 18 and older. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 7 to 35 with higher scores indicating greater severity of anxiety.
Time Frame: Baseline (T1), 1 month (T2), and 4 months (T3)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video Library Group | Flyer Library Group
Number analyzed (Participants) | 58 | 57
score on a scale
  PROMIS Anxiety Time 1 | 63.71 (8.34) | 63.86 (8.16)
  PROMIS Anxiety Time 2: number analyzed (Participants) | 52 | 49
  PROMIS Anxiety Time 2 | 62.66 (8.60) | 61.40 (7.88)
  PROMIS Anxiety Time 3: number analyzed (Participants) | 49 | 50
  PROMIS Anxiety Time 3 | 62.11 (8.66) | 59.99 (8.91)
Statistical Analysis 1: Comparison: Video Library Group vs Flyer Library Group; Test type: Superiority; p = 0.30, Regression, Linear

7. Secondary Outcome: PROMIS Life Satisfaction Scale T-Scores
Description: PROMIS (Patient-Reported Outcomes Measurement Information System) Life Satisfaction Short Form is a 5-item for that assesses one's cognitive evaluation of life experiences and whether one likes his/her life or not. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always). The raw scores are summed and converted to the corresponding T-Score. PROMIS uses T-scores with a population mean of 50 and a standard deviation of 10. A higher score represents more life satisfaction.
Time Frame: Baseline (T1), 1 month (T2), and 4 months (T3)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Video Library Group | Flyer Library Group
Number analyzed (Participants) | 58 | 57
T-Score
  PROMIS Life Satisfaction Time 1 | 40.56 (6.76) | 41.62 (6.77)
  PROMIS Life Satisfaction Time 2: number analyzed (Participants) | 51 | 48
  PROMIS Life Satisfaction Time 2 | 45.04 (9.80) | 47.78 (10.73)
  PROMIS Life Satisfaction Time 3: number analyzed (Participants) | 51 | 49
  PROMIS Life Satisfaction Time 3 | 46.13 (9.18) | 50.04 (9.47)
Statistical Analysis 1: Comparison: Video Library Group vs Flyer Library Group; Test type: Superiority; p = 0.06, Regression, Linear

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Video Library Group | Flyer Library Group
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/57
Other Adverse Events (participants affected / at risk) | 0/58 | 0/57

LIMITATIONS AND CAVEATS:
One of the outcomes Skill Score: Compromise, posed significant challenges during the roleplay and coding stages. We were not able to reflect the full complexity of this in the roleplay scenarios, which resulted in an overly simple scenario. Scores were consistently high across all time points and across both groups, meaning that we ran into a ceiling effect and did not see significant change.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2025-02-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT06281171/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT06281171/SAP_001.pdf
  • Informed Consent Form (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT06281171/ICF_002.pdf